CLINICAL TRIAL: NCT07202806
Title: A Study on the Application of Aromatherapy Combined With Transcranial Magnetic Stimulation in Insomnia of Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dandan Wu (Other)
Responsible Party: Sponsor-Investigator, Dandan Wu, Associate Professor, Second Affiliated Hospital of Nanchang University
Organization: Second Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024B1366
Record Dates: First submitted 2025-09-10; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcranial magnetic stimulation (No Intervention)
- Aromatherapy + transcranial magnetic stimulation (Experimental): Experimental:Aromatherapy + transcranial magnetic stimulation
  1.Aromatherapy is made from self-made sachet of traditional Chinese medicine.Its components (albizzia, Angelica dahurica, cardamom, Polygala, Evodia, Magnolia, Acorus calamus) are 10g each. Place the pillow 1 hour in advance. It is forbidden to play with your mobile phone or turn off the lights before going to bed.2.The r repetitive transcranial magnetic acupuncture apparatus produced by Jiangxi brain Control Technology Development Co., Ltd. is used and operated by professional therapists.Before treatment, the resting exercise threshold of each patient was tested: 10 pulse stimuli were given to find out the lowest stimulus intensity that could cause more than 50 microvolts.Parameter setting: 90% RMT 1Hz, each sequence lasts 12s, stimulation 10s, interval 2s. The treatment time was 20min/, once per day for 5 days per week, lasting for 3 weeks.
  Interventions: Behavioral: Aromatherapy

INTERVENTIONS:
Behavioral: Aromatherapy — 1.Aromatherapy is made from self-made sachet of traditional Chinese medicine.Its components (albizzia, Angelica dahurica, cardamom, Polygala, Evodia, Magnolia, Acorus calamus) are 10g each. Place the pillow 1 hour in advance. It is forbidden to play with your mobile phone or turn off the lights before going to bed.
  Arms: Aromatherapy + transcranial magnetic stimulation

SUMMARY:
Exploring the application efficacy of aromatherapy combined with transcranial magnetic stimulation on insomnia in patients with cerebral stroke

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* Insomnia patients
* Sign the informed consent form, cooperate voluntarily
* Accord with the diagnosis of "insomnia" in traditional Chinese medicine
* Evaluation has no taboo on transcranial magnetism
* The age range is between 24 and 65

Exclusion Criteria:

* Disturbance of consciousness
* Cognitive impairment
* Mental abnormality
* Sleep apnea syndrome
* Restless leg syndrome

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory sleep monitoring | From enrollment to the end of treatment for 3 weeks
  The average length of sleep in a week Sleep breathing monitoring was determined by evaluation before and after treatment. The main purpose of this study was to observe whether the average sleep time of patients increased significantly after treatment.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index,PSQI | From enrollment to the end of treatment for 3 weeks
  Pittsburgh sleep quality index（PSQI） The Pittsburgh Sleep quality Index (PSQI) was used to evaluate the sleep status of the patients before treatment and after three weeks of treatment. The total score of the scale was 0-21. The higher the score, the worse the sleep quality.